CLINICAL TRIAL: NCT04651465
Title: Norwegian Tuning in to Kids Effectivity Study
Acronym: N-TIK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Evalill Bølstad, PhD, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2020-11-13; First posted 2020-12-03 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Emotional Intelligence
Keywords: emotion socialization; intervention; Tuning in to Kids

STUDY DESIGN:
Intervention Model Description: Randomised control trial, where both intervention and control group participants are assessed at baseline, and then the intervention groups get the intervention, and all group participants are assessed at follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuning in to Kids parenting program (Experimental): Intervention groups receive the Tuning in to Kids parenting program
  Interventions: Behavioral: Tuning in to Kids
- Business as usual (No Intervention): control groups have "business as usual", and then get offered the intervention program after one year follow-up assessment.

INTERVENTIONS:
Behavioral: Tuning in to Kids — A parenting program that includes 6 group supervisions of parents, where emotion coaching and promotion of kids emotional competence are main focus.
  Arms: Tuning in to Kids parenting program

SUMMARY:
The current Randomised Controlled Trial study delivers and evaluate an evidence-based prevention program from Australia (Tuning in to Kids: TIK) to parent of preschool children. Reports from parents and preschool teachers are used to determine whether the program leads to universal benefits of improved wellbeing and reduced mental health difficulties for children and parents.

DETAILED DESCRIPTION:
The study recruits approximately 250 parents of preschool children through local kindergartens to evaluate the N-TIK program as a universal and selective prevention program. The study will use a cluster randomized controlled design and comparing an intervention with a wait-list control sample. Baseline measurement (Time 1) are gathered from parents, children and teachers and include measurement of parenting, parent functioning, child emotion competence, child behavior and child kindergarten adjustment. Following baseline assessment families is allocated into Intervention or Wait-list conditions. Intervention parents attend a 6-session group parenting program where they learn to emotion coach their children and regulate their own emotions. These groups are facilitated by selected research team facilitators. Post-program, Intervention parents complete program evaluation measures (Time 2) to provide program feedback. At 12-month follow-up (Time 3) baseline assessments are repeated for Intervention and Wait-list participants with preschool teachers reporting on children's adjustment. Wait-list parents are then offered the N-TIK program delivered by community practitioners who have been trained by the project team in the intervention and have previously co-facilitated groups alongside the research group facilitators. This ensures the program can be used beyond just the research study building sustainability of the preventive intervention in the municipalities

ELIGIBILITY:
Inclusion Criteria:

* Parent of a preschool child aged 4-5 years old

Exclusion Criteria:

* Under the age of 18
* Not able to read and write in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent Emotion Socialization Questionnaire (PESQ) | Up to 18 months
  Parent Emotion Socialization Questionnaire (PESQ) is a scale with items that are scored from 1 to 5, where 5 indicates high levels of specific parenting beliefs (i.e. emotion coaching and emotion dismissive beliefs). Change in PESQ from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.
Coping with children negative emotions scale (CCNES) | Uo to 18 months
  Coping with children negative emotions scale (CCNES) is a scale with items that are scored from 1 to 7, where 7 indicates high levels of specific parenting behavior (i.e. supportive and nonsupportive parenting behavior). Change in CCNES from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.
Eysenck's child behavior questionnaire (ECBI) | Up to 18 months
  Eysenck's child behavior questionnaire (ECBI) is a scale with items that are scored from 1 to 7, where 7 indicates high levels of behavior problems. Change in ECBI from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.
Preschool anxiety scale - revised (PAS-R) | Up to 18 months
  Preschool anxiety scale - revised (PAS-R) is a scale with items that are scored from 1 to 5, where higher score indicates higher levels of anxiety. Change in PAS-R from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.

SECONDARY OUTCOMES:
Affect Integration Inventory (AII) | Up to 18 months
  Affect Integration Inventory (AII) is a scale with scores from 0 to 8, where 8 indicates high affect integration. Change in AII from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.
Difficulties with Emotion Regulation Scale (DERS) | Up to 18 months
  Difficulties with Emotion Regulation Scale (DERS) is a scale with scores from 1 to 5, where 5 indicates more difficulties with emotion regulation. Change in DERS from baseline to post intervention (up to 6 months after baseline) to 1 year follow-up measured by questionnaire reports.

CONTACTS AND LOCATIONS:
Overall Officials: Evalill Bølstad, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway